CLINICAL TRIAL: NCT00909233
Title: LEVITRA® 20mg Special Drug Use Investigation (Long-term)
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Medical Director, Bayer Yakuhin Ltd
Other Study IDs: 13930; LV0701JP
Record Dates: First submitted 2009-05-08; First posted 2009-05-27 (Estimated); Last update posted 2014-12-15 (Estimated); Status verified 2014-12

CONDITIONS: Erectile Dysfunction
Keywords: Erectile dysfunction,; Phosphodiesterase Inhibitors
MeSH Terms: conditions — Erectile Dysfunction | interventions — Vardenafil Dihydrochloride

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Vardenafil, (Levitra, BAY38-9456)

INTERVENTIONS:
Drug: Vardenafil, (Levitra, BAY38-9456) — Patients under daily life treatment receiving Levitra according to local drug information.

SUMMARY:
This investigation targets either the patients of 18 years-old or older and under 65 years-old with organic or mixed erectile dysfunction (ED) who cannot obtain sufficient efficacy by dose 10mg of Levitra, and the target patients dose is increased to Levitra 20mg. This investigation will be limited to the patients whose tolerability of Levitra 10mg is judged to be no problem.

ELIGIBILITY:
Inclusion Criteria:

* This investigation targets either the patients of 18 years-old or older and under 65 years-old with organic or mixed erectile dysfunction who cannot obtain sufficient efficacy by dose 10mg of Levitra, and the target patients dose is increased to Levitra 20mg. This investigation will be limited to the patients whose tolerability of Levitra 10mg is judged to be no problem.

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 1221 (Actual)
Dates: Start 2007-08; Primary Completion 2010-03 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Efficacy of patients with LEVITRA treatment | After 6 months

SECONDARY OUTCOMES:
LEVITRA treatment improved the patient's erection | After 6 months
LEVITRA improved the patient's erection after Minimum and Maximum Intervals between LEVITRA intake and the start of intercourse | After 6 months
Reporting a second successful intercourse within 24 hours of dosing | After 6 months
Patients prefer LEVITRA over last Erectile Dysfunction treatment | After 6 months
Tolerability of patients with LEVITRA treatment | After 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Japan